CLINICAL TRIAL: NCT06442995
Title: Superiority Randomized Double-blind Controlled Trial of Epidural Magnesium Sulfate Addition Versus Placebo on the Occurrence of Acute Post-caesarean Urinary Retention
Brief Title: Evaluation of the Efficacy of the Addition of Magnesium Sulfate to Morphine on the Occurrence of Acute Urinary Retention Following Epidural Anesthesia for Cesarean Section.
Acronym: EPIMAG
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PO24038*
Record Dates: First submitted 2024-05-23; First posted 2024-06-05 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulfate (Experimental): Injection of 500 mg magnesium sulfate + 2 mg morphine into the epidural space
  Interventions: Drug: Injection of 500 mg magnesium sulfate + 2 mg morphine into the epidural space
- Isotonic saline (Placebo Comparator): Injection of Isotonic saline + 2 mg morphine into the epidural space
  Interventions: Drug: Injection of Isotonic saline + 2 mg morphine into the epidural space

INTERVENTIONS:
Drug: Injection of 500 mg magnesium sulfate + 2 mg morphine into the epidural space — When the patient agrees to enter the protocol, the investigators randomize the patient and proceed to the injection of morphine 2 mg into the epidural catheter + magnesium sulfate 500 mg
  Arms: Magnesium Sulfate
Drug: Injection of Isotonic saline + 2 mg morphine into the epidural space — When the patient agrees to enter the protocol, the investigators randomize the patient and proceed to Injection of morphine 2 mg into the epidural catheter + isotonic saline. This is the protocol the investigators use in daily practice for parturients who have undergone Caesarean section, in line with the French recommendations of anesthesia societies
  Arms: Isotonic saline

SUMMARY:
Peri-medullary anesthesia is the preferred anesthetic technique for Caesarean surgery. Compared with general anesthesia, it reduces maternal and fetal morbidity and mortality, as well as postoperative pain. However, this technique exposes the patient to the adverse effects of peri-medullary morphine, particularly the risk of postoperative urinary retention. Urinary retention during the first 72 hours after Caesarean section affects around 33% of parturients.

This is a particularly debilitating event for parturients, exposing them to the risk of further urinary catheterization, increased theoretical risk of urinary tract infection, traumatic urethral injury, hindered accelerated rehabilitation and altered maternal satisfaction.

Several studies have demonstrated the benefits of adding magnesium sulfate to epidural anesthesia for Caesarean sections, notably by reducing postoperative pain.

Magnesium sulfate may also have a facilitating effect on postoperative micturition, thanks to its sympathicolytic effect.

This hypothesis is supported by a retrospective study carried out in our maternity hospital, which showed a 15% reduction in post-Caesarean urinary retention when women were given magnesium sulfate in addition to the drugs traditionally used for epidurals.

This little-known property needs to be clarified

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the efficacy of the addition of epidural magnesium sulfate in reducing the occurrence of acute post-Caesarean urine retention.

In fact, the incidence of acute urine retention after epidural anaesthesia for Caesarean section is around 33%. Two encouraging studies suggest that adding magnesium sulfate to epidurals could reduce the incidence of acute urine retention by 15%.

This study will be carried out on the obstetric population of the REIMS maternity hospital, starting in summer 2024. It is a randomized, double-blind, placebo-controlled clinical trial. The number of subjects required is calculated at 290 patients, with a power of 80% and an alpha risk of 5%. The statistical hypothesis is that magnesium sulfate reduces the incidence of acute urine retention by 15% compared with placebo (isotonic saline).

Parturients will be informed of the study during a pre-anaesthetic consultation in the 6th month of pregnancy.

Some of these patients will be scheduled for delivery by caesarean section. The remaining patients will be scheduled for a vaginal delivery, which may end up being an emergency caesarean section (10-15% of patients).

After the Caesarean section, patients are taken to the post-procedure monitoring room, where they are monitored for 2 hours.

It is at this point that patients are examined to verify the inclusion and non-inclusion criteria of the protocol. If the inclusion and non-inclusion criteria are met, our teams will provide patients with explanatory documents on our protocol, as well as a consent form for their signature.

When the patient agrees to enter the protocol, the investigators randomize her to one of the following groups:

* Group A: injection of morphine 2 mg into the epidural catheter + magnesium sulfate 500 mg
* Group B: injection of morphine 2 mg into the epidural catheter + isotonic saline.

Group B is the control group. This is the protocol we use in daily practice for parturients who have undergone Caesarean section, in line with the French recommendations of anesthesia societies.

This reduces the parturient's postoperative pain for 20-24 hours. Group A will be the experimental group. Patients will be monitored in the post-natal care unit for 72 hours. The investigators will carry out the same monitoring and care as a parturient outside the protocol. Various data on diuresis, the quantity of urine in the bladder visualized by ultrasound, and the need for urinary catheterization will be recorded.

Statistical analyses will determine whether the incidence of acute urine retention differs between each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone scheduled or emergency Caesarean section surgery under extended epidural anesthesia or combined epidural and spinal anesthesia at the Reims University Hospital.
* Patients who have just undergone caesarean section and have the epidural catheter in place in the post-interventional monitoring room (SSPI).
* Patients who agree to take part in the research and have signed the informed consent form
* Patients of legal age
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Minor patients
* Patients protected by law
* Patients allergic to local anesthetics, morphine or magnesium sulfate
* Patients with severe renal insufficiency (GFR < 30 ml/min)
* Patients with pre-pregnancy mictional disorders
* Patients with an American Society of Anesthesiologists (ASA) score of 4
* Patients undergoing caesarean section under general anaesthesia, after failure of perimedullary anaesthesia
* Patients with accidental intraoperative injury to the urinary tract
* Patients who have received intravenous magnesium sulfate in the 24 hours preceding cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
diuresis | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided